CLINICAL TRIAL: NCT00276172
Title: An Open-Label, Multicenter Extension Study to Evaluate the Safety and Tolerability of Natalizumab in Subjects With Multiple Sclerosis Who Have Completed Studies C-1801, C-1802, or C-1803
Brief Title: Open-Label Natalizumab Safety Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-1808
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natalizumab (Experimental): Open-label natalizumab
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Natalizumab 300 mg by IV infusion, every 4 weeks, for up to 24 months
  Other Names: Tysabri

SUMMARY:
The primary objective of this study is to determine the safety and the immunogenicity of extended treatment with natalizumab when administered at a dose of 300 mg intravenously (IV) to subjects with multiple sclerosis (MS) who have completed natalizumab Studies C-1801, C-1802, or C-1803.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent.
* Must be an MS subject who has completed natalizumab Study C-1801, C-1802 or C-1803

Exclusion Criteria:

* History of, or available abnormal laboratory results, indicative of any significant disease that would preclude treatment.
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity
* A clinically significant infectious illness within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1615 (Actual)
Dates: Start 2003-12; Primary Completion 2005-10 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
The safety endpoints under consideration will be the incidence of adverse events, changes in laboratory evaluations, vital signs, and physical examinations. The incidence of development of antibodies to natalizumab will also be assessed. | Month 24

SECONDARY OUTCOMES:
EDSS scores and assessments of relapse. | Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Michael Panzara, MD, MPH, Study Director — Biogen; Paul O'Connor, MD, Principal Investigator — Unity Health Toronto; Eve Versage, Study Chair — Biogen Idec. Contact for more details
Locations (1):
- Performed at only C-1801, C-1802, and C-1803 sites globally. No general public enrollment. Biogen Idec is located in, Cambridge, Massachusetts, United States